CLINICAL TRIAL: NCT03745625
Title: A Single-center, Open-label, Randomized, Double-crossover, Propofol-controlled, Two-stage Study Evaluating the Safety and Pharmacokinetics/Pharmacodynamics of IV Maintenance Dose After An Initial Dose and IV Single Loade Dose Plus Maintenance Dose of HSK3486 Emulsion fo Injection in Healthy Subjects
Brief Title: A Study Evaluating the Safety and Pharmacokinetics/Pharmacodynamics of HSK3486
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-102
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): First-stage: 1mg/kg/h, 0.4mg/kg/h; Second-stage:Single loading dose: 0.2mg/kg, maintenance dose: 0.35mg/kg/h,
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): First-stage: 5mg/kg/h, 2mg/kg/h; Second-stage:Single load ing dose: 1mg/kg, maintenance dose: 1.75mg/kg/h
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — First-stage:after an initial dose of 1mg/kg/h, If the BIS is in the range of 80 to 60 and the continuous RASS score = 3 or one time RASS score ≤ -4, the 0.4 mg/kg/h maintenance dose is administered. The total infusion time was 4h.
  Second-stage: a single loading dose of 0.2 mg/kg given over 1 minute, then a continuous infusion of maintenance dose 0.35 mg/kg/h for a total infusion time of 12h.
  Arms: HSK3486
Drug: Propofol — First-stage: after an initial dose of 5mg/kg/h, If the BIS is in the range of 80 to 60 and the continuous RASS score = 3 or one time RASS score ≤ -4, the 0.4 mg/kg/h maintenance dose is administered. The total infusion time was 4h.
  Second-stage: loading dose of 1mg/kg given over 1 minute, then a continuous infusion of maintenance dose 1.75 mg/kg/h for a total infusion time of 12h.
  Arms: Propofol

SUMMARY:
This is a Phase I, single-center, open-label, randomized,two-way crossover, propofol-controlled, two-stage study evaluating the safety and pharmacokinetics/pharmacodynamics of IV maintenance dose after an initial dose and IV single loade dose plus maintenance dose of HSK3486 emulsion for injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females with full capacity for civil conduct, aged ≥ 18 and ≤ 49 years old;
2. Body weight > 45 kg, and body mass index (BMI) ≥ 19 and ≤26 kg/m2;
3. Blood pressure between 90-140/60-90 mmHg; heart rate between 60-99 bpm; body temperature between 35.8-37.5 °C; respiration rate between 12-20 breaths per minute; SpO2 when inhaling > 95%;
4. Normal physical examinations, laboratory examinations (routine blood test, blood biochemistry and routine urinalysis), and 12-Lead ECG, or abnormal but without clinical significance; no potential difficult airway (modified Mallampati score I-III);
5. No previous history of major organ primary diseases, such as liver, kidneys, digestive tract, blood, and metabolic diseases; no history of malignant hyperthermia and other genetic conditions; no history of mental/neurological diseases; No history of epilepsy; no contraindications for deep sedation/general anesthesia; no clinically significant history of anesthesia accidents;
6. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with trial protocol.

Exclusion Criteria:

1. Known sensitivity to propofol, excipients in propofol medium-/long-chain triglyceride emulsion injection, excipients in HSK3486 emulsion injection (soybean oil, glycerin, triglyceride, egg lecithin, sodium oleate, and sodium hydroxide); history of drug allergies (including anesthetics), allergic diseases, or those with hyperactive immune response;
2. History of drug abuse or any signs of chronic benzodiazepines use (such as insomnia, anxiety, spasms) within 3 months prior to screening, or a positive urine drug test during screening;
3. Participated in clinical trials involving any medications or medical devices within 3 months prior to screening, or subjects who have participated in 3 or more drug clinical trials within the past year;
4. Serious infection, trauma or major surgery within 4 weeks before screening; or acute disease with clinical significance (determined by the investigator) within 2 weeks before screening, including GI diseases or infections (such as respiratory or CNS infections);
5. In receipt of propofol, other sedatives/anesthetics and/or opioid analgesics or compounds containing analgesics within 3 days prior to screening;
6. In receipt of prescription drugs, Chinese herbal medicines, over-the-counter drugs or food supplements (such as vitamins and calcium supplements) other than contraceptives, paracetamol, oral non-steroidal anti-inflammatory drugs, topical over-the-counter preparations, within 2 weeks prior to enrollment; unless the principal investigator (PI) and the sponsor agree that the medication has no effect on the safety and PK/PD results of the trial;
7. History of cardiovascular diseases such as: postural hypotension, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, tachycardia/bradycardia requiring medication, third-degree atrioventricular block or QTcF interval ≥ 450 ms (Fridericia's correction formula);
8. Impaired respiratory function, history of obstructive pulmonary disease, history of asthma, sleep apnea syndromes; history of failed tracheal intubation; history of bronchospasm requiring treatment within 3 months prior to screening; acute upper respiratory tract infection, and with obvious symptoms such as fever, wheezing, nasal congestion and cough within 1 week prior to baseline;
9. History of GI tract diseases: Gastrointestinal obstruction, active GI bleed, potential for reflux and aspiration;
10. Laboratory results that meet any of the following during screening/enrollment:

    * Positive test for either HBsAg, HCV, HIV, or syphilis;
    * Abnormal hepatic or renal function confirmed after re-examination;

      * ALT or AST > 1×ULN;
      * Creatinine > 1×ULN;
      * TBIL > 1.5×ULN;
11. History of alcohol abuse within 3 months prior to screening, abuse defined as average of > 2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive blood alcohol concentration during screening;
12. Blood donation or blood loss ≥ 200 mL within 30 days before the trial; plasma donation or plasma exchange within 7 days before the trial;
13. Subjects who continue to smoke, drink alcohol, or consume any food or beverages containing xanthine or caffeine, to participate in strenuous physical activities and other factors that may affect drug absorption, distribution, metabolism, and excretion within 2 days prior to enrollment; subjects who are unable to fast for 6 hours prior to dose administration;
14. Subjects expected to have surgery or hospitalization during the trial;
15. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 1 month after the completion of the trial (including male subjects);
16. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
blood pressure（systolic, diastolic and mean arterial pressure） | from the screening to 3 days post-dose
  safety endpoits
heart rate | from the screening to 3 days post-dose
  safety endpoits
respiratory rate | from the screening to 3 days post-dose
  safety endpoits
blood oxygen saturation | from the screening to 3 days post-dose
  safety endpoits
Number of patients with adverse events | from the baseline to 3 days post-dose
  safety endpoits

SECONDARY OUTCOMES:
Richmond Agitation Sedation Scale( scores：+4~-5) | -30 minutes before administration until the subject is completely awakened post administration on day 1
  Change from baseline in Richmond Agitation Sedation Scale(RASS) score
Bispectral index | -30 minutes before administration until the subject is completely awakened post administration on day 1
Sedation/anesthesia satisfaction, satisfaction assessment of subjects, anesthesiologists, and endoscopic physicians | -30 minutes before administration until the subject is completely awakened post administration on day 1
Terminal elimination half life | -30 minutes before administration until 24 hours post administration on day 1
Total clearance | -30 minutes before administration until 24 hours post administration on day 1
Volume of distribution | -30 minutes before administration until 24 hours post administration on day 1
plasma concentration at the end of infusion | -30 minutes before administration until 24 hours post administration on day 1

OTHER OUTCOMES:
area under curve from time 0 to the last measurable blood sampling time (AUC0-last) | -30 minutes before administration until 24 hours post administration on day 1
area under curve from time 0 to infinite time (AUC0-inf) | -30 minutes before administration until 24 hours post administration on day 1
Peak concentration | -30 minutes before administration until 24 hours post administration on day 1
time to peak observed (Tmax) | -30 minutes before administration until 24 hours post administration on day 1

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, China